CLINICAL TRIAL: NCT04446390
Title: Evaluation of Remineralization Potential of Preventive Regimens Containing Herbal-based Compared to Fluoride-based Toothpastes in High Caries Risk Patients With Initial Carious Lesions: Randomized Clinical Trial
Brief Title: Preventive Regimens With Herbal and Fluoride Toothpaste on Remineralization in High Caries Patients With Initial Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yomna Hussin, Master degree studnet, Conservative Dentistry Department, Faculty of Dentistry, Cairo University., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Himalaya herbal toothpaste
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preventive regimen using Herbal toothpaste(Himalaya) (Experimental): The regimen includes herbal toothpaste containing "Neem , Miswak , Babool and Pomegranate" (Himalaya Complete Care). Chew xylitol gum 2 pieces four times per day for 5 minutes after meals.
  Interventions: Other: Himalaya complete care toothpaste
- preventive regimen using Fluoride based toothpaste(colgate) (Active Comparator): preventive regimen using Fluoride based toothpaste (colgate cavity protection). Participants will be using a fluoride-based toothpaste (colgate cavity protection), (1450 ppm Sodium monofluorophosphate). chew xylitol gum 2 pieces four times per day for 5 minutes after meals.
  Interventions: Other: colgate cavity protection

INTERVENTIONS:
Other: Himalaya complete care toothpaste — Herbal toothpaste as a part of a caries preventive regimen
  Arms: preventive regimen using Herbal toothpaste(Himalaya)
Other: colgate cavity protection — fluoride toothpaste as a part of a caries preventive regimen
  Arms: preventive regimen using Fluoride based toothpaste(colgate)

SUMMARY:
This study will be conducted to assess the effect of different preventive regimens using herbal toothpaste versus fluoride toothpaste on the management of remineralization and caries risk in high caries risk patients.

DETAILED DESCRIPTION:
Dental caries is a major universal health problem with multiple etiological factors, so looking for economical and accurate plans for recognizing high-risk persons, and multiple risk factors to reduce the risk, in addition to caries management, using a caries risk assessment to detect the person who will develop caries, and provide them with suitable preventive and treatment regimens to disruption the disease procedure.

The treatment should evade invasive treatments and a large emphasis on prevention (using fluoride toothpaste, solutions, patient education, and so on), to achieve the aim of new dentistry (minimal intervention). The application of such a regimen to manage initial caries lesions allows the dentist to reverse initial lesions with the minimal victim of healthy dental tissues.

ELIGIBILITY:
* Inclusion criteria of the participants:

  1. Healthy patients with free medical history.
  2. Age range 15-50 years.
  3. Patients with high caries risk assessment according to Cariogram.
  4. Patients with initial carious lesions at the facial surface of any teeth
  5. High plaque index
  6. Not under antibiotic therapy either at the time of the study or up to the last month before the start of the study
* Exclusion criteria of the participants:

  1. Patients with a compromised medical history.
  2. Patients with dentin caries
  3. Extreme plaque accumulation and periodontal problems
  4. Completely edentulous patients
  5. Participants with a history of allergy to any of the drugs or chemicals used in the study.
  6. Patients on any antibiotics during the past month
* Inclusion criteria of the teeth:

  1. The WSLs with LF measurements inside the range 14-20 were involved in this study.
  2. The lesions with scoring either 2 or 3 according to (ICDAS) scoring were included in the study
* Exclusion criteria of the teeth:

  1. The white spot lesion scoring is (<14) or (>20) according to diagnodent
  2. The white spot lesion scoring is other than 2, 3 according to ICDAS
  3. White spot lesions due to hypomineralization or fluorosis

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Remineralization of initial carious lesions | Outcomes will be evaluated at baseline, after 1 week, after 4 weeks and after 12 weeks.
  changes in fluorescence of white spot lesions will be evaluated after reminerlization by using Diagnodent scoring (0-20): healthy teeth (0-14), initial carious lesions (14-20), dentinal caries (more than 20)

SECONDARY OUTCOMES:
Caries risk assessment | Outcomes will be evaluated at baseline, after 1 week, after 4 weeks and after 12 weeks.
  Change in caries risk assessment by "cariogram software" as each patient data is collected in order to be inserted into the "Cariogram software" which in turn will evaluate this data and lead to a pie chart showing the chance of avoiding new caries as percentage.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Cairo University, Faculty of Oral and Dental Medicine, Cairo
  - Cairo University, Cairo